CLINICAL TRIAL: NCT00817388
Title: Correlating Ic/Pbs Symptoms With Urine Biomarkers
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Michael Chancellor, MD, Beaumont Hospitals
Other Study IDs: 2008-294
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-06

CONDITIONS: Interstitial Cystitis; Pelvic Pain
Keywords: Interstitial cystitis; pelvic pain
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Urine specimen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients will be asked to provide a urine specimen and complete a questionnaire.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Completion of a brief survey tool and providing an urine specimen. The study purpose is to improve our understanding of interstitial cystitis and painful pelvic syndrome.

DETAILED DESCRIPTION:
The purpose of the study is to improve our understanding of the IC/PBS and develop new treatments. Participation in the study will allow us to compare clinical information, obtained by completion of a brief survey, with substances found in the a urine specimen that is donated to the Beaumont Biobank.

ELIGIBILITY:
Inclusion:

1. Men and women with interstitial cystitis/painful bladder syndrome greater than 18 years old
2. Male and female controls without a history of IC/PBS diagnosis

Exclusion:

1. Unable to complete questionnaires and/or give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with and without intersitial cystitis/painful pelvic pain will be asked to provide an urine specimen and complete a brief questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To correlate IC/PBS symptoms with urine biomarkers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chancellor, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States